CLINICAL TRIAL: NCT06386549
Title: Effect of a Tele-rehabilitation Programme in Children With Burns: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LIAO Peng (Other)
Responsible Party: Sponsor-Investigator, LIAO Peng, Mr., The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20220424001
Record Dates: First submitted 2024-03-25; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Burns; Tele-rehabilitation; Scar; Children
Keywords: tele-rehabilitation; parental stress; scar management; quality of life
MeSH Terms: conditions — Burns; Cicatrix | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tele-rehabilitation (Experimental): experimental group received an 12-week tele-rehabilitation program, which included face-to-face access to silicone pads, pressure garments, splint and other tools necessary for burn recovery. The tele-rehabilitation program was used for intervention and regular follow-up.
  Interventions: Behavioral: tele-rehabilitation
- routine post-discharge rehabilitation (Active Comparator): The control group also received an 12-week follow-up, but only on the basis of face-to-face access to silicone pads, pressure garments, splint and other tools necessary for burn recovery.
  Interventions: Behavioral: tele-rehabilitation

INTERVENTIONS:
Behavioral: tele-rehabilitation — Using the social networking tool WeChat, families of children with burns are educated and trained through texts, photos, voice messages, and live videos, twice a week for a total of 12 weeks

SUMMARY:
The goal of this clinical trial is to compare tele-rehabilitation and routine post-discharge rehabilitation in children with burn injuries. The main questions it aims to answer are:

* Is tele-rehabilitation better for improving the quality and outcomes of care for burn children?
* Is tele-rehabilitation more effective in improving scar management in children with burns injuries?
* Is tele-rehabilitation more effective in improving perceived stress in parents of children with burns injuries?

DETAILED DESCRIPTION:
In this study, experimental group received a 12-week tele-rehabilitation program, which included face-to-face access to silicone pads, pressure garments, splint and other tools necessary for burn recovery. The tele-rehabilitation program was used for intervention and regular follow-up.

The control group also received a 12-week follow-up, but only on the basis of face-to-face access to silicone pads, pressure garments, splint and other tools necessary for burn recovery.

Researchers will compare whether the trial group has better the quality and outcomes of care and scarring for children and parents who perceived stress.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are based on the recommendations of the American Burn Association.
* Child suffered from burn injury 3-6 years old and had survived the burn event.
* The burn severity quantified by the total body surface area（TBSA）burned is equal or more than 1%.
* TBSA burned is the estimated proportion of the body with second or third degree burns.
* Burns involving neck, trunk，limbs and face.
* Only Chinese parents will be recruited.

Exclusion Criteria:

* 1.Insufficient parental Chinese language proficiency required to complete questionnaires.
* Parents cannot use social software (such as WeChat, QQ, etc.) for video, picture, and text communication after discharge.
* The main caregiver is someone other than the parents.
* Children did not live at home with their parents, such as hospitalization, boarding school, etc.
* Children who are receiving rehabilitation treatment.
* Children who have other severe disease, like cerebral palsy.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The scars of children with burns | baseline , 4 weeks, 8 weeks, and 12 weeks (post-test)
  Ultrasound assessment of scar thickness, The DermaLab Combo assessment of scar Transepidermal Water Loss (TEWL), pigmentation, hydration and elasticity.
  The normal skin thickness is about 0.07-1.2mm, while the thickness of hypertrophic scars increases with the severity.
  The DermaLab Combo® (Cortex Technologies, Denmark) is a commercially available skin testing device. It is a high-specification device based on proven technologies. It is an easy to use and commercially available device, making it a viable option for scar assessment in both clinical and research settings.
  The worse the scar condition, the greater the Transepidermal Water Loss (TEWL), the darker the pigmentation (the larger the value), the smaller the hydration, and the smaller the elasticity (the larger the value).
The quality and outcomes of care for burn children | baseline , 4 weeks, 8 weeks, and 12 weeks (post-test)
  The health outcomes burn questionnaire (HOBQ) for infants and children 6 years of age and younger is developed by American Burn Association/Shriners Hospitals for Children.
  The HOBQ has a total of 55 items, calculated on a hundred-point scale, the higher the score, the better. Consists of 10 subscale, and each item is also converted into a percentage system. For the same score, the higher the better. There are 5 items for play, 4 items for language, 7 items for fine motor skills, 7 items for gross motor skills, 9 items for behavior, 5 items for family, 7 items for pain/itching, 3 items for appearance, 5 items for satisfaction, and 3 items for concern/worry. The number of items per scale ranges from two to nine. All subscales relate to the past month,except the subscale 'satisfaction'. The questionnaire has been translated into Chinese, and the reliability and validity of its Chinese version have also been confirmed.

SECONDARY OUTCOMES:
psychological stress of caregvers | baseline , 4 weeks, 8 weeks, and 12 weeks (post-test)
  The Perceived Stress Scale (PSS) is the world's most widely used instrument to measure perceived stress, 14 items，its Chinese version is widely used and has good reliability and validity. Each item in the PSS questionnaire is rated on a five-point Likert scale, ranging from 0 (never) to 4 (very often). Participants are asked to indicate the frequency with which they have experienced each event over the past month.The total score on the PSS can range from 0 to 56. Higher scores indicate a higher level of perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Shumei, Study Chair
Locations (1):
- Hongkong Poly Uiniversity, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/49/NCT06386549/ICF_000.pdf